CLINICAL TRIAL: NCT06684639
Title: An Open Clinical Study on the Safety and Efficacy of Autologous GD2-CAR T Cells in the Treatment of Relapsed Refractory Neuroblastoma
Brief Title: A Study on the Efficacy of GD2-CAR T Cells in the Treatment of Neuroblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yihai2024
Record Dates: First submitted 2024-08-28; First posted 2024-11-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Relapsed; Refractory
MeSH Terms: conditions — Neuroblastoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): GD2 positive relapsed or refractory neuroblastoma
  Interventions: Biological: GD2-CAR-T cell

INTERVENTIONS:
Biological: GD2-CAR-T cell — Split intravenous infusion of GD2-CAR-T cells [dose escalating infusion of (1-100)x10^6 GD2-CAR-T cells/kg]

SUMMARY:
Neuroblastoma (NB) is a malignant tumor of the sympathetic nervous system.Chemotherapy and autologous hematopoietic stem cell transplantation are the main treatments for neuroblastoma, and the prognosis of patients with high-risk recurrence and refractory treatment is very poor. There is a large unmet medical need in patients with relapsed refractory neuroblastoma, and further research into new therapeutic approaches is needed for these patients.GD2 is a dissialic ganglioside expressed by neuroectodermal tumors. The proportion of GD2 expression in neuroblastoma is up to 100%, so GD2 is a specific target for neuroblastoma immunotherapy and an ideal target for CAR-T treatment of neuroblastoma.

DETAILED DESCRIPTION:
The subjects received the target dose of GD2-CAR-T from 1×106 to 1×108 /kg. Each subject will start with a low dose of 1×106/kg and if there are no significant side effects will be increased to the next dose until the maximum tolerated dose is reached. A variety of adverse events (including neurological events, hematological events, infections, and secondary tumors) will be collected from the time of infusion of CAR T cells to 24 months after infusion. To understand the complete response rate (CR) and partial response rate (PR) at 3 months; Recurrence rate, progression-free survival (PFS) and overall survival (OS) after 1 to 5 years of GD2-CAR-T reinfusion; The amount and duration of GD2-CAR-T in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. All cases were diagnosed as neuroblastoma with positive expression of GD2 antigen in tumor cells. Informed consent of patient or guardian.
2. Diagnosis of recurrent/refractory neuroblastoma.
3. At least 2 weeks or 5 half-lives (whichever is shorter) from the beginning of preconditioning chemotherapy after prior systemic treatment.
4. Toxic reactions caused by previous antitumor therapy must be stabilized and restored to ≤ grade 1.
5. Over 1 years old, under 18 years old.
6. Physical strength score 0-3 (ECOG standard).
7. No obvious active infection.
8. Expected survival ≥3 months
9. Adequate kidney, liver, lung and heart function, defined as creatinine clearance (estimated by the Cockcroft Gault formula) > 60 mL/min; Serum ALT/AST ≤ 2.5 ULN; Total bilirubin ≤1.5 ULN, excluding subjects with Gilbert's syndrome; Cardiac ejection fraction ≥ 50%, echocardiography confirmed centropericardial effusion, and ECG showed no clinically significant abnormal findings. There was no clinically significant pleural effusion. Baseline blood oxygen saturation under indoor ventilation was > 92%.
10. The serum pregnancy test results of fertile women must be negative (women who have undergone surgical sterilization or at least 2 years after menopause are considered to be infertile).

Exclusion Criteria:

1. The subject has had other malignancies, non-melanoma skin tumors, carcinoma in situ (e.g. Cervix, bladder, breast), unless disease-free survival of at least 3 years.
2. There is an uncontrollable infection, including fungal, bacterial, viral or other.
3. Known human immunodeficiency virus (HIV) infection.
4. Known history of hepatitis B (HBsAg positive) or hepatitis C (HCV antibody positive). Subjects with latent or prehepatitis B infection (defined as HBcAb positive and HBsAg negative) can be enrolled only if PCR tests for HBV DNA are negative. In addition, these subjects were required to undergo a monthly PCR test for HBV DNA. Participants who are serologically positive for HCV antibodies can also be enrolled if their PCR test results for HCV RNA are negative.
5. Existing or past CNS disease, such as seizures, cerebrovascular ischemia/bleeding, dementia, cerebellar disease, or any CNS-related autoimmune disease.
6. Serious heart disease, such as uncontrolled or symptomatic arrhythmia, congestive heart failure, or myocardial infarction within 6 months prior to screening, or any grade 3 (moderate) or 4 (severe) heart disease (according to the New York Heart Society Functional Grading Method NYHA).
7. A history of myocardial infarction, angioplasty or stent placement, unstable angina pectoris, or other clinically significant heart disease in the 12 months prior to enrollment.
8. Any medical condition that may affect the evaluation of safety or efficacy.
9. Have had severe rapid hypersensitivity reactions to any of the drugs to be used in this study.
10. Live vaccine should be administered within ≤6 weeks before starting the pretreatment regimen.
11. Pregnant or lactating female subjects.
12. Male or female subjects who do not consent to effective contraception from the time they sign informed consent until 6 months after completing immune cell therapy.
13. Subjects judged by the investigator had difficulty in completing all visits or procedures required by the study protocol (including follow-up visits), or were not compliant enough to participate in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 24 months
  Adverse events are evaluated with CTCAE V4.03
Overall response rate (ORR) | 24 months
  ORR includes CR, PR,MR.SD,PD.Complete response (CR)#All components CR.Partial response (PR)#PR in at least one component and all other components CR,minimal disease (bone marrow), PR or not involved at baseline.Minor response (MR)#PR or CR in at least one component but at least one other component with SD; no component with PD.Stable disease (SD)#SD in one component with no better than SD or not involved at baseline in any other component, no component with PD.Progressive disease (PD)#Any component with PD.

SECONDARY OUTCOMES:
Duration of overall response (DOR) | 24 months
  Duration of overall response will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Progression-free survival(PFS) | 24 months
  PFS will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Overall survival(OS) | 24 months
  OS will be assessed from the CAR-T cell infusion to death or last follow-up.

OTHER OUTCOMES:
The duration of CAR T-cells in vivo | 24 months
  The time of CAR-T cells' persistence in blood and the copies of CAR-T cells
CAR-T related cytokine expression | 24 months
  CAR-T related cytokine expression.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Yi, Ph.D, Principal Investigator — The General Hospital of Western Theater Command
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No